CLINICAL TRIAL: NCT05008653
Title: Surveying Nutrient Assessment With Photographs of Meals (SNAPMe) Study
Acronym: SNAPMe
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1730621
Record Dates: First submitted 2021-06-28; First posted 2021-08-17 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Food Characteristics
Keywords: Artificial intelligence; Dietary records; Food systems; Computer science; Sustainability; Nutrition

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SnapMe Study is a single-group, prospective study that requires healthy adults to maintain food diaries in order to develop benchmark data for the prediction of food characteristics.

DETAILED DESCRIPTION:
The purpose of this study is to develop a method that uses photography to accurately calculate the types and amounts of nutrients in meals that are consumed by healthy participants, thereby replacing the use of electronic food records. Researchers expect about 100 healthy individuals at UC Davis and around the U.S. will join to participate in this research. Participation in this study will involve taking pictures of every meal and snack the individual consumes using a smartphone for 3 days (2 weekdays, 1 weekend day) and uploading the images to a mobile phone application called Bitesnap. In addition, the participant will be asked to complete online food records on the same days using the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24-2020). Each participant will have 4 weeks to complete the study. The study website can be viewed here: https://snapme.ucdavis.edu/

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults
2. Has a social security number or Tax ID
3. Age 18-65 years of age
4. Lives anywhere in the United States of America
5. Has been weight-stable (has not lost or gained 10% of body weight) within the past 3 months
6. Currently owns a smart phone (Android or iPhone)
7. Has owned and used a smart phone for at least 12 months
8. Consumes at least 3 meals per day
9. Consumes at least 50% of meals that are prepared at/from home vs. outside the home (dine-in restaurants, take-out, etc.)
10. Prepares at least 50% of the prepared meals within their household
11. Willingness to refrain from participating in any experimental trials during this study period
12. Willingness to refrain from having any non-emergency, elective surgeries during the study period
13. Willingness to eat different/variety of foods for each meal over the three days of dietary record collection
14. Willingness to refrain from consuming meal substitution items (examples: Slimfast shake, Soylent, meal replacement bars) over the three days of dietary record collection
15. Willingness to download and use an app linked to their smart phone's camera and photo storage
16. Willingness to spend 1-2 hours per day on each of the three study days to: 1)enter detailed information about each meal they consume using an online record system and an app on their smart phone and 2) take and upload photos of their meals on their smart phone
17. Willingness to refrain from sharing meals with other participants during data collection
18. Passes a food matching test on the online screening survey with score >70%.

Exclusion Criteria:

1. Currently pregnant or plans to become pregnant several weeks prior to enrollment and during the study period
2. History of any type of eating disorder (anorexia nervosa, bulimia, etc.)
3. Use of restrictive diets such as caloric restriction or intermittent fasting of more than 12 hours that has resulted in weight loss greater than 10% of their body weight within the past 3months ordiets
4. Anyone the investigator feels is not an applicable participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults living anywhere in the United States of America between the ages of 18 and 65.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
Primary Study Endpoint | 3 days
  Construct a library with thousands of meals and snacks and images of these meals and snacks.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCullough ML. Dietary assessment in the digital age: the ongoing quest for better methods. Am J Clin Nutr. 2018 Jan 1;107(1):1-2. doi: 10.1093/ajcn/nqx066. No abstract available. PMID 29381804
- [Background] Timon CM, van den Barg R, Blain RJ, Kehoe L, Evans K, Walton J, Flynn A, Gibney ER. A review of the design and validation of web- and computer-based 24-h dietary recall tools. Nutr Res Rev. 2016 Dec;29(2):268-280. doi: 10.1017/S0954422416000172. PMID 27955721
- [Background] Subar AF, Kipnis V, Troiano RP, Midthune D, Schoeller DA, Bingham S, Sharbaugh CO, Trabulsi J, Runswick S, Ballard-Barbash R, Sunshine J, Schatzkin A. Using intake biomarkers to evaluate the extent of dietary misreporting in a large sample of adults: the OPEN study. Am J Epidemiol. 2003 Jul 1;158(1):1-13. doi: 10.1093/aje/kwg092. PMID 12835280